CLINICAL TRIAL: NCT00937287
Title: Understanding HPV Vaccination Among Rural African American Primary Caregivers and Daughters
Brief Title: Human Papilloma Virus (HPV) Vaccination Among Rural African American Primary Caregivers and Daughters
Status: Completed | Type: Observational
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Steve Kogan, Principal Investigator, University of Georgia
Other Study IDs: MISP 36701
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Human Papillomavirus
Keywords: HPV; African American; Rural

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- youth and caregivers
  Interventions: Other: There is no intervention in this study.

INTERVENTIONS:
Other: There is no intervention in this study. — No intervention is provided in this study as it is exploratory.

SUMMARY:
African American women living in the rural South are twice as likely as Caucasian women to develop cervical cancer and die of invasive cervical cancer at a higher rate than any other racial/ethnic group in the US (1). Reasons for low HPV vaccination rates among rural African Americans are not well understood. HPV vaccination compliance is likely influenced by barriers to health care access, misinformation regarding vaccinations, religious beliefs related to sexual health and behaviors, and mistrust of the medical community (2, 3). Because the vaccination of minors requires primary caregiver consent, vaccination commitment and compliance is strongly influenced by family beliefs and communication regarding health and sexuality. To date, little research has examined the cultural, familial, and intrapersonal influences on HPV vaccination compliance among rural African American women. This study will address these gaps in the literature and provide data needed to develop effective interventions and health promotion materials to encourage HPV vaccination among rural African American women.

From a pool of approximately 800 families who are participating in ongoing longitudinal research through the Center for Family Research at the University of Georgia, the investigators will recruit 200 rural female African American youth aged 13-17 who have not received the HPV vaccine and their primary caregivers (n=200) into an observational, prospective study on vaccination commitment and compliance. The investigators hypotheses are as follows:

1. Sociocultural factors that rural African Americans experience, including discrimination, previous health care experience, religious beliefs, and community norms regarding HPV vaccination and adolescent sexual behavior, will forecast primary caregivers' HPV vaccination commitment and compliance for their daughters. The investigators also predict that primary caregivers' HPV-related knowledge and attitudes will mediate this association.
2. Sociocultural factors will influence sexual health-related family communication and interaction, primary caregivers' and youths' HPV-related attitudes, and HPV vaccination commitment and compliance.
3. Primary caregivers' attitudes, youths' attitudes, and family health communication will contribute to youths' and caregivers' vaccination commitment and compliance.
4. Youths' sexual behavior will influence their attitudes, family health communication, and vaccination commitment and compliance.

ELIGIBILITY:
Inclusion Criteria:

* Rural African American girls aged 13-17
* Female parent or primary caregiver of participating daughter

Exclusion Criteria:

* Girls can not be younger than age 13, or older than 17
* The target's female parent or primary caregiver must also live in the same household and agree to participate

Ages: 13 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The sample will include rural, female African American youth aged 13-17 (n=200) and their primary caregivers (n=200) who reside in the same household.
Sampling Method: Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2009-07; Primary Completion 2011-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
HPV vaccination compliance | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie R. Burwell, PhD, Principal Investigator — University of Georgia
Locations (1):
- The Center for Family Research, Athens, Georgia, United States

REFERENCES:
- [Background] Saraiya M, Ahmed F, Krishnan S, Richards TB, Unger ER, Lawson HW. Cervical cancer incidence in a prevaccine era in the United States, 1998-2002. Obstet Gynecol. 2007 Feb;109(2 Pt 1):360-70. doi: 10.1097/01.AOG.0000254165.92653.e8. PMID 17267837
- [Background] Brewer NT, Fazekas KI. Predictors of HPV vaccine acceptability: a theory-informed, systematic review. Prev Med. 2007 Aug-Sep;45(2-3):107-14. doi: 10.1016/j.ypmed.2007.05.013. Epub 2007 Jun 2. PMID 17628649
- [Background] Cates JR, Brewer NT, Fazekas KI, Mitchell CE, Smith JS. Racial differences in HPV knowledge, HPV vaccine acceptability, and related beliefs among rural, southern women. J Rural Health. 2009 Winter;25(1):93-7. doi: 10.1111/j.1748-0361.2009.00204.x. PMID 19166567